CLINICAL TRIAL: NCT03317171
Title: Studio Monocentrico in Doppio Cieco Randomizzato Dell'Effetto di Una Miscela di Flavonoidi ed Acidi Grassi Naturali in Pazienti Affetti da Distrofia Muscolare
Brief Title: Safety and Efficacy of a Flavonoids- and omega3s-based Compound for the Treatment of Muscular Dystrophies
Acronym: PRO1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1768
Record Dates: First submitted 2017-10-11; First posted 2017-10-23 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Muscular Dystrophies; Muscle Inflammation
Keywords: dietary supplementation; flavonoids; omega 3
MeSH Terms: conditions — Muscular Dystrophies; Myositis, Inclusion Body | interventions — Flavonoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated group (Experimental): oral administration of flavonoids, DHA and EPA, once a day for 24 weeks.
  Interventions: Dietary Supplement: Flavonoids, DHA, EPA
- Placebo group (Placebo Comparator): oral administration of placebo compound, once a day for 24 weeks.
  Interventions: Dietary Supplement: placebo compound

INTERVENTIONS:
Dietary Supplement: Flavonoids, DHA, EPA — oral administration
  Arms: Treated group
Dietary Supplement: placebo compound — oral administration
  Arms: Placebo group

SUMMARY:
The study aimed to assess the safety and, partially, the efficacy of dietary supplementation of a flavonoids-, DHA- and EPA-based natural supplement in non-ambulant DMD boys and in a cohort of LGMD and FSHD patients to compare its effect in MDs of different aetiology and to eventually highlight any differences in inflammatory involved pathways. To assess safety, patient's laboratory parameters were monitored and adverse events recorded, while efficacy was evaluated through performance scale questionnaire and strength measurement (6 minute walking test and Biodex System 4 Dynamometer parameter evaluation). This study was conceived as proof of principle for the safe use of flavonoids/omega3s-based compound as an adjuvant in the management of neuromuscular disorders; besides, its efficacy in alleviating symptoms linked to secondary effects of genetic mutation as inflammation, muscular pain and weakness was assessed.

ELIGIBILITY:
INCLUSION CRITERIA

* documented genetic and histological diagnosis of DMD, FSHD and LGMD;
* absence of severe cardiac and pulmonary disease;
* age superior to 9 years for DMD, between 9 and 70 years for LGMD and between 20 and 70 years for FSHD;
* glucocorticosteroid treatment for 6 or more months (stable dose and regimen for ≥3 months before screening) and for the duration of the study;
* adhesion to inform consent by same patients or parents/tutors for minors.

EXCLUSION CRITERIA

* severe cardiac and pulmonary disease;
* positive hepatitis B surface antigen (HBsAg) test, positive hepatitis C and HIV tests;
* low kidney and liver functionality;
* autoimmune disorders;
* mental retardation (IQ via Wechsler Intelligence Scale < 70);
* psychological-psychiatric disorders; adverse psychosocial conditions;
* known allergies to some of compounds to be used in the trial;
* pathologies occurring just before or during the trial (fever, metabolic disorders, drug abuse);
* enrollment to other trials (steroids regime won't be considered in this list)

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — males, for patients affected by Duchenne muscular dystrophy
Enrollment: 29 (Actual)
Dates: Start 2016-02-28 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Safety of the administered supplements | month 0 and month +6
  blood tests, to monitor any possible change before and after the study
Safety of the administered supplements | month 0 and month +6
  ECG, to monitor any possible change before and after the study
Safety of the administered supplements | month 0 and month +6
  neurological clinical assessment, to monitor any possible change before and after the study

SECONDARY OUTCOMES:
Efficacy outcome - functional changes after the treatment | month 0 and month +6
  Biodex System 4 Dynamometer for quantitative measures (muscle strength and resistance)
Efficacy outcome - functional changes after the treatment | month 0 and month +6
  6 Minute Walking Test for quantitative measures (muscle strength and resistance)
Efficacy outcome - functional changes after the treatment | month 0, month +2, month +4, month +6
  EK (Egen Klassifikation) scale to assess funtionality of patients with significative impairments. Min. score: 0 - max. score 30
Efficacy outcome - functional changes after the treatment | month 0, month +2, month +4, month +6
  ACTIVLIM (Activity Limitation) scale. The scale measures activity limitations for patients with upper and/or lower limb impairments and has been validated in patients affected by neuromuscular disorders. Min. score: 0 - max. score 36
Efficacy outcome - functional changes after the treatment | month 0, month +2, month +4, month +6
  ABILHAND (manual ability for adults with upper limb impairments) scale. The scale measures manual ability for adults with upper limb impairments.Min. score: 0 - max. score 36

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Derived] Sitzia C, Meregalli M, Belicchi M, Farini A, Arosio M, Bestetti D, Villa C, Valenti L, Brambilla P, Torrente Y. Preliminary Evidences of Safety and Efficacy of Flavonoids- and Omega 3-Based Compound for Muscular Dystrophies Treatment: A Randomized Double-Blind Placebo Controlled Pilot Clinical Trial. Front Neurol. 2019 Jul 23;10:755. doi: 10.3389/fneur.2019.00755. eCollection 2019. PMID 31396142